CLINICAL TRIAL: NCT01566305
Title: The Effects of Buttermilk With or Without Lutein-enriched Egg Yolk on the Serum LDL Cholesterol Concentration of Slightly Hypercholesterolaemic Volunteers
Brief Title: Effects of Buttermilk on Serum LDL Cholesterol Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL33461.068.10
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Hypercholesterolemia; Buttermilk; Dietary Modification; Cardiovascular Disease
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — Buttermilk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Buttermilk with added egg yolk (Experimental)
  Interventions: Dietary Supplement: Buttermilk with added egg yolk
- Buttermilk without added egg-yolk (Experimental)
  Interventions: Dietary Supplement: Buttermilk without added egg-yolk
- Skimmed milk with added egg-yolk (Experimental)
  Interventions: Dietary Supplement: Skimmed milk with added egg-yolk
- Skimmed milk without added egg yolk (Placebo Comparator)
  Interventions: Dietary Supplement: Skimmed milk without added egg yolk

INTERVENTIONS:
Dietary Supplement: Buttermilk without added egg-yolk — Buttermilk without added egg-yolk
  Arms: Buttermilk without added egg-yolk
Dietary Supplement: Buttermilk with added egg yolk — Buttermilk with added egg yolk
  Arms: Buttermilk with added egg yolk
Dietary Supplement: Skimmed milk with added egg-yolk — Skimmed milk with added egg-yolk
  Arms: Skimmed milk with added egg-yolk
Dietary Supplement: Skimmed milk without added egg yolk — Skimmed milk without added egg yolk
  Arms: Skimmed milk without added egg yolk

SUMMARY:
Rationale and objective:

Based on the results of a pilot study, the objective of the present study is to evaluate whether buttermilk lower serum LDL cholesterol concentrations and can prevent the serum LDL cholesterol raising effects of eggs.

Study Design:

The study has a randomized placebo-controlled factorial 2x2 design. The total study duration is 14 weeks, consisting of a 2 weeks run-in period and a 12 weeks experimental period. Subjects will be stratified for age, gender and BMI over the experimental groups.

Study population:

One hundred and eight healthy male and female subjects, aged 18-70 years, with slightly elevated serum total cholesterol concentrations (5.5-8.0 mmol/l).

Intervention:

During the entire study period, volunteers are instructed to consume a diet according to the Dutch dietary guidelines (35 en% fat (10 en% saturated fat), 50-55 en% carbohydrates). During the two weeks run-in period all subjects will drink daily at lunch 100 mL skimmed milk. During the 12 weeks experimental period, a first group of subjects will continue drinking the skimmed milk (control group), while a second group will consume a low-fat buttermilk, a third group skimmed milk enriched with egg-yolk, and a fourth group egg-yolk incorporated into a low-fat buttermilk based beverage. The egg-yolk will be enriched in lutein. Whole egg consumption (others than provided by us) is not allowed during the entire study.

Main study parameters/endpoints:

Measurements will be performed during the run-in period (days 0, 11 and 14) and during the experimental period (days 56, 95 and 98). The main effects (egg-yolk and buttermilk consumption) will be calculated as the absolute differences between values obtained at the end of the experimental (average days 95 and 98) and run-in (average days 11 and 14) periods. The primary endpoint is the change in serum LDL cholesterol concentrations. Secondary endpoints are changes in serum total and HDL cholesterol, triacylglycerol, apoA-I, apoB and hsCRP concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years
* Fasting serum total cholesterol between 5.5 - 8.0 mmol/l
* Fasting plasma glucose < 7.0 mmol/l
* BMI between 25-30 kg/m2
* non-smoking
* Willingness to abstain for the duration of the study from egg consumption

Exclusion Criteria:

* unstable body weight (weight gain or loss >3 kg in the past 3 months)
* allergic for eggs or egg-rich products
* allergic or intolerant for cow-milk (lactose) based products
* indication for treatment with cholesterol-lowering drugs according to the Dutch Cholesterol Consensus
* use of medication or a diet known to affect serum lipid or glucose metabolism - active cardiovascular disease (for instance congestive heart failure) or recent (<6 months) event, such as acute myocardial infarction or cerebro-vascular accident
* not willing to stop the consumption of vitamin supplements, fish oil capsules or products rich in plant stanol or sterol esters 3 weeks before the start of the study
* men: consumption of >21 alcohol consumptions a week
* women: consumption of >14 alcohol consumptions a week
* abuse of drugs
* pregnant or breastfeeding women
* participation in another biomedical study within 1 month prior to the screening visit
* having donated blood (as blood donor) within 1 month prior to the screening visit or planning to do so during the study
* impossible or difficult venipuncture as evidenced during the screening visits

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2012-05-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
Change in serum LDL cholesterol concentrations | LDL cholesterol will be measured at day 0, 11, 14, 56, 95 and 98 during the study

SECONDARY OUTCOMES:
Changes in serum total and HDL cholesterol, triacylglycerol, apoA-I, apoB and hsCRP concentrations | Serum total and HDL cholesterol, triacylglycerol, apoA-I and ApoB will be measured at day 0, 11, 14, 56, 95 and 98 during the study. hsCRP concentrations will be measured at day 11, 14, 95 and 98.

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Severins N, Mensink RP, Plat J. Effects of lutein-enriched egg yolk in buttermilk or skimmed milk on serum lipids & lipoproteins of mildly hypercholesterolemic subjects. Nutr Metab Cardiovasc Dis. 2015 Feb;25(2):210-7. doi: 10.1016/j.numecd.2014.10.003. Epub 2014 Oct 13. PMID 25456153
- See also: Related Info — https://doi.org/10.1016/j.numecd.2014.10.003